CLINICAL TRIAL: NCT00172978
Title: Indications and Related Factors for Caesarean Delivery, 1996 to 2002.
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700346
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-10-27 (Estimated); Status verified 2005-04

CONDITIONS: Labor

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To study the effect of elective pain relief analgesia in labor on mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

- women in labor

Exclusion Criteria:

* women with special conditions

Ages: 10 Years to 60 Years | Sex: Female
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Lin Hwa, MD, Principal Investigator
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan